CLINICAL TRIAL: NCT00284271
Title: Feasibility and Efficacy of BACOPP-21 for Patients > 60 Years With Intermediate or Advanced Hodgkins Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BACOPP-21
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Hodgkin´s Lymphoma
Keywords: Hodgkin´s Lymphoma; eldery patients; primary diagnosis
MeSH Terms: interventions — Cyclophosphamide; Prednisone; Vincristine; Bleomycin

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Adramycin
Drug: Procarbacine
Drug: Prednisone
Drug: Vincristine
Drug: Bleomycin
Drug: Erythropoietin beta

SUMMARY:
This study is designed to test (1) feasibility and efficiancy of new BACOPP regimen and (2) toxicity, overall response and FFTF.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin´s lymphoma (histologically proven)
* CS (PS) I and II with one of the risk factors a-d

  1. bulky mediastinal mass (> 1/3 maximum transverse thorax diameter)
  2. extranodal involvement
  3. ESR > 50 (A), > 30 (B-symptoms)
  4. 3 or more lymph node areas involved
* CS (PS) III and IV
* Written informed consent

Exclusion Criteria:

* Leukocytes <3000/microl
* Platelets <100000/microl
* Hodgkin´s Disease as "composite lymphoma"
* Activity index (WHO) < grade 2

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Josting, Dr., Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

REFERENCES:
- [Result] Halbsguth TV, Nogova L, Mueller H, Sieniawski M, Eichenauer DA, Schober T, Nisters-Backes H, Borchmann P, Diehl V, Engert A, Josting A. Phase 2 study of BACOPP (bleomycin, adriamycin, cyclophosphamide, vincristine, procarbazine, and prednisone) in older patients with Hodgkin lymphoma: a report from the German Hodgkin Study Group (GHSG). Blood. 2010 Sep 23;116(12):2026-32. doi: 10.1182/blood-2009-11-253211. Epub 2010 Jun 15. PMID 20551376